CLINICAL TRIAL: NCT06779916
Title: Study of the Autophagy/Apoptosis Balance in Placental Vascular Pathologies
Brief Title: Autophagy/Apoptosis Balance in Placental Vascular Pathologies
Acronym: GROSSAUTOP-2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2024-1/SB01
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Complications; Pre-Eclampsia; Growth Retardation, Intrauterine
Keywords: trophoblasts; autophagy; apoptosis; placenta; pregnancy
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia; Fetal Growth Retardation | interventions — Hematologic Tests; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A biobank (plasmabank, serum bank, mononuclear cells) will be set up for ancillary studies on other markers of placental vascular pathologies and venous thromboembolic disease.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women developing placental vascular complications: Pregnant adult women developing placental vascular complications such as preeclampsia and/or intrauterine growth retardation, hospitalized and delivering at Nimes University Hospital.
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Urine test

INTERVENTIONS:
Diagnostic Test: Blood test — 16 blood samples (16 tubes, i.e. 55.3 ml) will be taken at inclusion. Pregnant women will be seen every month as part of their pregnancy follow-up, and blood (11 tubes, i.e. 35.5 ml) and urine samples will be taken at each follow-up visit.
  At delivery, a systematic blood sample will be taken as part of the usual care, and an additional 11 tubes of blood (35.5 ml) will be taken.
Diagnostic Test: Urine test — Urine samples will be taken at the inclusion visit and at each follow-up visit.

SUMMARY:
Pregnancy increases the risk of thrombosis. Placenta-mediated diseases are a risk factor for cardiovascular pathologies and can lead to maternal-fetal morbidity and mortality. It is essential to understand the cellular and molecular mechanisms of dysfunctions at the vascular-placental interface so that systemic vascular risk can be characterized and, ultimately, screened for, on the basis of new markers (targeted preventive management).

Deregulated autophagy could be the starting point for cell death by apoptosis or necrosis leading to complications.

The pathophysiological mechanisms involved in trophoblast apoptosis are incompletely described. This project follows on from the GrossAuTop-1 study, which investigated the intra- and inter-individual variability of autophagy and apoptosis activities in women during pregnancy. The aim of this project is to study autophagy and apoptosis activities specifically in women developing a placental vascular complication during pregnancy.

DETAILED DESCRIPTION:
Pregnancy increases the risk of thrombosis. Diseases mediated by the placenta are a risk factor for cardiovascular pathologies. They are responsible for significant maternal-fetal morbidity and mortality. Understanding and exploring the cellular and molecular mechanisms of dysfunctions at the vascular-placental interface could provide arguments for understanding systemic vascular risk, characterizing it and ultimately screening for it on the basis of new markers, thus paving the way for targeted preventive management, feeding into the general principle of precision medicine.

Autophagy enables cell development, differentiation and survival, but if deregulated, it could be the starting point for cell death by apoptosis or necrosis, and promote the development of complications.

The pathophysiological mechanisms involved in trophoblast apoptosis are incompletely described. A deregulation of the trophoblast proliferation/cell death balance could be at the origin of placental pathologies. The regulation of autophagy and autophagy-dependent events during pregnancy have not been fully identified.

We hypothesize that there is an intratrophoblastic dialogue between autophagy and apoptosis mechanisms, with the promotion of one partially inhibiting the other. The increase in trophoblastic autophagy during pregnancy could thus constitute an anti-apoptosis defense phenomenon, whose depletion would lead to cellular apoptosis and pathogenic consequences when it devastates the syncytiotrophoblast.

This project follows on from the GrossAuTop-1 study, which investigated the intra- and inter-individual variability of autophagy and apoptosis activities in women during pregnancy: the inclusions corresponded to all-pregnant women, the majority of whom developed a normal pregnancy. The aim of this project is to study autophagy and apoptosis activities specifically in women developing a placental vascular complication during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women developing a placental vascular complication (preeclampsia and/or intrauterine growth retardation), hospitalized and delivering at Nimes University Hospital.
* Pregnant woman with free and informed consent.
* Pregnant woman affiliated with and/or benefiting from a health insurance scheme.

Exclusion criteria:

* Multiple pregnancy.
* Presence of hypertension and/or proteinuria prior to pregnancy.
* Participant in an interventional drug study.
* Persons in a period of exclusion determined by another study.
* Persons under court protection, guardianship or curatorship.
* Persons unable to give consent.
* Persons for whom it is impossible to give informed information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: An initial analysis of the data will make it possible to describe the population.
  Quantitative variables will be expressed as mean and standard deviation, or median and quartiles. Qualitative variables will be expressed in headcount and percentage.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein | Baseline
  Level of autophagy in trophoblastic test cells quantified by the percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein
Percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein | Month 1
  Level of autophagy in trophoblastic test cells quantified by the percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein
Percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein | Month 2
  Level of autophagy in trophoblastic test cells quantified by the percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein
Percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein | Month 3
  Level of autophagy in trophoblastic test cells quantified by the percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein
Percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein | Month 4
  Level of autophagy in trophoblastic test cells quantified by the percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein
Percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein | At delivery
  Level of autophagy in trophoblastic test cells quantified by the percentage of cells expressing LC3 (microtubule-associated protein light chain 3) protein

SECONDARY OUTCOMES:
Apoptosis activity | Baseline
  Percentage of cells expressing annexin-V in pregnant women developing placental vascular pathology
A. Apoptosis activity | Month 1
  Percentage of cells expressing annexin-V in pregnant women developing placental vascular pathology
A. Apoptosis activity | Month 2
  Percentage of cells expressing annexin-V in pregnant women developing placental vascular pathology
A. Apoptosis activity | Month 3
  Percentage of cells expressing annexin-V in pregnant women developing placental vascular pathology
A. Apoptosis activity | Month 4
  Percentage of cells expressing annexin-V in pregnant women developing placental vascular pathology
A. Apoptosis activity | At delivery
  Percentage of cells expressing annexin-V in pregnant women developing placental vascular pathology
B. Autophagy/apoptosis balance | Baseline
  Ratio between percentage of cells expressing LC3 protein and percentage of cells expressing annexin-V
B. Autophagy/apoptosis balance | Month 1
  Ratio between percentage of cells expressing LC3 protein and percentage of cells expressing annexin-V
B. Autophagy/apoptosis balance | Month 2
  Ratio between percentage of cells expressing LC3 protein and percentage of cells expressing annexin-V
B. Autophagy/apoptosis balance | Month 3
  Ratio between percentage of cells expressing LC3 protein and percentage of cells expressing annexin-V
B. Autophagy/apoptosis balance | Month 4
  Ratio between percentage of cells expressing LC3 protein and percentage of cells expressing annexin-V
B. Autophagy/apoptosis balance | At delivery
  Ratio between percentage of cells expressing LC3 protein and percentage of cells expressing annexin-V
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: LC3 protein | Baseline
  LC3 protein will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: LC3 protein | Month 1
  LC3 protein will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: LC3 protein | Month 2
  LC3 protein will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: LC3 protein | Month 3
  LC3 protein will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: LC3 protein | Month 4
  LC3 protein will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: LC3 protein | At delivery
  LC3 protein will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: cells expressing annexin-V | Baseline
  Cells expressing annexin-V will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: cells expressing annexin-V | Month 1
  Cells expressing annexin-V will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: cells expressing annexin-V | Month 2
  Cells expressing annexin-V will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: cells expressing annexin-V | Month 3
  Cells expressing annexin-V will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: cells expressing annexin-V | Month 4
  Cells expressing annexin-V will be measured as a %
C.Kinetics of different biological activities (autophagy, apoptosis, autophagy/apoptosis balance) during pregnancy follow-up: cells expressing annexin-V | At delivery
  Cells expressing annexin-V will be measured as a %
D. Concentration of circulating Placental Growth Factor | Baseline
  Circulating Placental Growth Factor measured on blood samples in pg/mL
D. Concentration of circulating Placental Growth Factor | Month 1
  Circulating Placental Growth Factor measured on blood samples in pg/mL
D. Concentration of circulating Placental Growth Factor | Month 2
  Circulating Placental Growth Factor measured on blood samples in pg/mL
D. Concentration of circulating Placental Growth Factor | Month 3
  Circulating Placental Growth Factor measured on blood samples in pg/mL
D. Concentration of circulating Placental Growth Factor | Month 4
  Circulating Placental Growth Factor measured on blood samples in pg/mL
D. Concentration of circulating Placental Growth Factor | At delivery
  Circulating Placental Growth Factor measured on blood samples in pg/mL
D. Concentration of circulating soluble fms-like tyrosine kinase receptor-1 | Baseline
  Circulating soluble fms-like tyrosine kinase receptor-1 measured on blood samples in pg/mL
D. Concentration of circulating soluble fms-like tyrosine kinase receptor-1 | Month 1
  Circulating soluble fms-like tyrosine kinase receptor-1 measured on blood samples in pg/mL
D. Concentration of circulating soluble fms-like tyrosine kinase receptor-1 | Month 2
  Circulating soluble fms-like tyrosine kinase receptor-1 measured on blood samples in pg/mL
D. Concentration of circulating soluble fms-like tyrosine kinase receptor-1 | Month 3
  Circulating soluble fms-like tyrosine kinase receptor-1 measured on blood samples in pg/mL
D. Concentration of circulating soluble fms-like tyrosine kinase receptor-1 | Month 4
  Circulating soluble fms-like tyrosine kinase receptor-1 measured on blood samples in pg/mL
D. Concentration of circulating soluble fms-like tyrosine kinase receptor-1 | At delivery
  Circulating soluble fms-like tyrosine kinase receptor-1 measured on blood samples in pg/mL
E. Correlation between autophagy/apoptosis balance and markers of renal function: proteinuria | Baseline
  Proteinuria will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: proteinuria | Month 1
  Proteinuria will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: proteinuria | Month 2
  Proteinuria will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: proteinuria | Month 3
  Proteinuria will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: proteinuria | Month 4
  Proteinuria will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: proteinuria | At delivery
  Proteinuria will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: creatinuria | Baseline
  Creatinuria will be measured in mmol/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: creatinuria | Month 1
  Creatinuria will be measured in mmol/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: creatinuria | Month 2
  Creatinuria will be measured in mmol/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: creatinuria | Month 3
  Creatinuria will be measured in mmol/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: creatinuria | Month 4
  Creatinuria will be measured in mmol/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: creatinuria | At delivery
  Creatinuria will be measured in mmol/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: C-reactive protein | Baseline
  C-reactive protein will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: C-reactive protein | Month 1
  C-reactive protein will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: C-reactive protein | Month 2
  C-reactive protein will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: C-reactive protein | Month 3
  C-reactive protein will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: C-reactive protein | Month 4
  C-reactive protein will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: C-reactive protein | At delivery
  C-reactive protein will be measured in mg/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: Fibrinogen | Baseline
  Fibrinogen will be measured in g/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: Fibrinogen | Month 1
  Fibrinogen will be measured in g/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: Fibrinogen | Month 2
  Fibrinogen will be measured in g/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: Fibrinogen | Month 3
  Fibrinogen will be measured in g/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: Fibrinogen | Month 4
  Fibrinogen will be measured in g/L
E. Correlation between autophagy/apoptosis balance and markers of renal function: Fibrinogen | At delivery
  Fibrinogen will be measured in g/L
E. Coagulation parameters : activated partial thromboplastin time | Baseline
  Activated partial thromboplastin time will be measured in seconds
E. Coagulation parameters : activated partial thromboplastin time | Month 1
  Activated partial thromboplastin time will be measured in seconds
E. Coagulation parameters : activated partial thromboplastin time | Month 2
  Activated partial thromboplastin time will be measured in seconds
E. Coagulation parameters : activated partial thromboplastin time | Month 3
  Activated partial thromboplastin time will be measured in seconds
E. Coagulation parameters : activated partial thromboplastin time | Month 4
  Activated partial thromboplastin time will be measured in seconds
E. Coagulation parameters : activated partial thromboplastin time | At delivery
  Activated partial thromboplastin time will be measured in seconds
E. Coagulation parameters : Prothrombin time | Baseline
  Prothrombin time will be measured in seconds
E. Coagulation parameters : Prothrombin time | Month 1
  Prothrombin time will be measured in seconds
E. Coagulation parameters : Prothrombin time | Month 2
  Prothrombin time will be measured in seconds
E. Coagulation parameters : Prothrombin time | Month 3
  Prothrombin time will be measured in seconds
E. Coagulation parameters : Prothrombin time | Month 4
  Prothrombin time will be measured in seconds
E. Coagulation parameters : Prothrombin time | At delivery
  Prothrombin time will be measured in seconds
E. Coagulation parameters : Fibrinogen | Baseline
  Fibrinogen will be measured in g/L
E. Coagulation parameters : Fibrinogen | Month 1
  Fibrinogen will be measured in g/L
E. Coagulation parameters : Fibrinogen | Month 2
  Fibrinogen will be measured in g/L
E. Coagulation parameters : Fibrinogen | Month 3
  Fibrinogen will be measured in g/L
E. Coagulation parameters : Fibrinogen | Month 4
  Fibrinogen will be measured in g/L
E. Coagulation parameters : Fibrinogen | At delivery
  Fibrinogen will be measured in g/L
E. Coagulation parameters : D-dimers | Baseline
  D-dimers will be measured in ng/mL
E. Coagulation parameters : D-dimers | Month 1
  D-dimers will be measured in ng/mL
E. Coagulation parameters : D-dimers | Month 2
  D-dimers will be measured in ng/mL
E. Coagulation parameters : D-dimers | Month 3
  D-dimers will be measured in ng/mL
E. Coagulation parameters : D-dimers | Month 4
  D-dimers will be measured in ng/mL
E. Coagulation parameters : D-dimers | At delivery
  D-dimers will be measured in ng/mL
E. Coagulation parameters : Fibrin monomers | Baseline
  Fibrin monomers will be measured in mg/mL
E. Coagulation parameters : Fibrin monomers | Month 1
  Fibrin monomers will be measured in mg/mL
E. Coagulation parameters : Fibrin monomers | Month 2
  Fibrin monomers will be measured in mg/mL
E. Coagulation parameters : Fibrin monomers | Month 3
  Fibrin monomers will be measured in mg/mL
E. Coagulation parameters : Fibrin monomers | Month 4
  Fibrin monomers will be measured in mg/mL
E. Coagulation parameters : Fibrin monomers | At delivery
  Fibrin monomers will be measured in mg/mL
E. Coagulation parameters : Thrombin generation time | Baseline
  Thrombin generation time will be measured in seconds
E. Coagulation parameters : Thrombin generation time | Month 1
  Thrombin generation time will be measured in seconds
E. Coagulation parameters : Thrombin generation time | Month 2
  Thrombin generation time will be measured in seconds
E. Coagulation parameters : Thrombin generation time | Month 3
  Thrombin generation time will be measured in seconds
E. Coagulation parameters : Thrombin generation time | Month 4
  Thrombin generation time will be measured in seconds
E. Coagulation parameters : Thrombin generation time | At delivery
  Thrombin generation time will be measured in seconds
Complete Blood Count : White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils | Baseline
  White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils will be measured in 10^9/L
Complete Blood Count : White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils | Month 1
  White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils will be measured in 10^9/L
Complete Blood Count : White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils | Month 2
  White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils will be measured in 10^9/L
Complete Blood Count : White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils | Month 3
  White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils will be measured in 10^9/L
Complete Blood Count : White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils | Month 4
  White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils will be measured in 10^9/L
Complete Blood Count : White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils | At delivery
  White blood cells, Lymphocytes, Neutrophils, Monocytes, Eosinophils and Basophils will be measured in 10^9/L
Complete Blood Count : Red blood cells | Baseline
  Red blood cells will be measured in 10^12/L
Complete Blood Count : Red blood cells | Month 1
  Red blood cells will be measured in 10^12/L
Complete Blood Count : Red blood cells | Month 2
  Red blood cells will be measured in 10^12/L
Complete Blood Count : Red blood cells | Month 3
  Red blood cells will be measured in 10^12/L
Complete Blood Count : Red blood cells | Month 4
  Red blood cells will be measured in 10^12/L
Complete Blood Count : Red blood cells | At delivery
  Red blood cells will be measured in 10^12/L
Complete Blood Count : Hemoglobin | Baseline
  Hemoglobin will be measured in g/L
Complete Blood Count : Hemoglobin | Month 1
  Hemoglobin will be measured in g/L
Complete Blood Count : Hemoglobin | Month 2
  Hemoglobin will be measured in g/L
Complete Blood Count : Hemoglobin | Month 3
  Hemoglobin will be measured in g/L
Complete Blood Count : Hemoglobin | Month 4
  Hemoglobin will be measured in g/L
Complete Blood Count : Hemoglobin | At delivery
  Hemoglobin will be measured in g/L
Complete Blood Count : Platelets | Baseline
  Platelets will be measured in %
Complete Blood Count : Platelets | Month 1
  Platelets will be measured in %
Complete Blood Count : Platelets | Month 2
  Platelets will be measured in %
Complete Blood Count : Platelets | Month 3
  Platelets will be measured in %
Complete Blood Count : Platelets | Month 4
  Platelets will be measured in %
Complete Blood Count : Platelets | At delivery
  Platelets will be measured in %
Complete Blood Count : Hematocrit | Baseline
  Hematocrit will be measured in %
Complete Blood Count : Hematocrit | Month 1
  Hematocrit will be measured in %
Complete Blood Count : Hematocrit | Month 2
  Hematocrit will be measured in %
Complete Blood Count : Hematocrit | Month 3
  Hematocrit will be measured in %
Complete Blood Count : Hematocrit | Month 4
  Hematocrit will be measured in %
Complete Blood Count : Hematocrit | At delivery
  Hematocrit will be measured in %
Complete Blood Count : Mean Corpuscular Volume | Baseline
  Mean Corpuscular Volume will be measured in f/L
Complete Blood Count : Mean Corpuscular Volume | Month 1
  Mean Corpuscular Volume will be measured in f/L
Complete Blood Count : Mean Corpuscular Volume | Month 2
  Mean Corpuscular Volume will be measured in f/L
Complete Blood Count : Mean Corpuscular Volume | Month 3
  Mean Corpuscular Volume will be measured in f/L
Complete Blood Count : Mean Corpuscular Volume | Month 4
  Mean Corpuscular Volume will be measured in f/L
Complete Blood Count : Mean Corpuscular Volume | At delivery
  Mean Corpuscular Volume will be measured in f/L
Complete Blood Count : Mean Corpuscular Hemoglobin | Baseline
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count : Mean Corpuscular Hemoglobin | Month 1
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count : Mean Corpuscular Hemoglobin | Month 2
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count : Mean Corpuscular Hemoglobin | Month 3
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count : Mean Corpuscular Hemoglobin | Month 4
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count : Mean Corpuscular Hemoglobin Concentration | Baseline
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count : Mean Corpuscular Hemoglobin Concentration | Month 1
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count : Mean Corpuscular Hemoglobin Concentration | Month 2
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count : Mean Corpuscular Hemoglobin Concentration | Month 3
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count : Mean Corpuscular Hemoglobin Concentration | At delivery
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Ferritin | Baseline
  Ferritin will be measured in ng/mL
Ferritin | Month 1
  Ferritin will be measured in ng/mL
Ferritin | Month 2
  Ferritin will be measured in ng/mL
Ferritin | Month 3
  Ferritin will be measured in ng/mL
Ferritin | Month 4
  Ferritin will be measured in ng/mL
Ferritin | At delivery
  Ferritin will be measured in ng/mL
F. Association between autophagy/apoptosis balance and the presence of constitutive thrombophilia | Baseline
  Constitutive thrombophilia: presence of prothrombin or factor V Leiden gene mutation, protein S, C, antithrombin deficiency will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of constitutive thrombophilia | Month 1
  Constitutive thrombophilia: presence of prothrombin or factor V Leiden gene mutation, protein S, C, antithrombin deficiency will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of constitutive thrombophilia | Month 2
  Constitutive thrombophilia: presence of prothrombin or factor V Leiden gene mutation, protein S, C, antithrombin deficiency will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of constitutive thrombophilia | Month 3
  Constitutive thrombophilia: presence of prothrombin or factor V Leiden gene mutation, protein S, C, antithrombin deficiency will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of constitutive thrombophilia | Month 4
  Constitutive thrombophilia: presence of prothrombin or factor V Leiden gene mutation, protein S, C, antithrombin deficiency will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of constitutive thrombophilia | At delivery
  Constitutive thrombophilia: presence of prothrombin or factor V Leiden gene mutation, protein S, C, antithrombin deficiency will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of acquired thrombophilia | Baseline
  Acquired thrombophilia: presence of anti-phospholipid antibodies (lupus anticoagulant and/or anti-b2-glycoprotein 1 and/or anti-cardiolipid) will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of acquired thrombophilia | Month 1
  Acquired thrombophilia: presence of anti-phospholipid antibodies (lupus anticoagulant and/or anti-b2-glycoprotein1 and/or anti-cardiolipid) will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of acquired thrombophilia | Month 2
  Acquired thrombophilia: presence of anti-phospholipid antibodies (lupus anticoagulant and/or anti-b2-glycoprotein1 and/or anti-cardiolipid) will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of acquired thrombophilia | Month 3
  Acquired thrombophilia: presence of anti-phospholipid antibodies (lupus anticoagulant and/or anti-b2-glycoprotein 1 and/or anti-cardiolipid) will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of acquired thrombophilia | Month 4
  Acquired thrombophilia: presence of anti-phospholipid antibodies (lupus anticoagulant and/or anti-b2-glycoprotein 1 and/or anti-cardiolipid) will be sought: YES/NO
F. Association between autophagy/apoptosis balance and the presence of acquired thrombophilia | At delivery
  Acquired thrombophilia: presence of anti-phospholipid antibodies (lupus anticoagulant and/or anti-b2-glycoprotein 1 and/or anti-cardiolipid) will be sought: YES/NO
Comparison of results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance | Baseline
  The results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance) will be compared with data obtained from the first GrossAuTop-1 study (normal pregnancy).
Comparison of results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance | Month 1
  The results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance) will be compared with data obtained from the first GrossAuTop-1 study (normal pregnancy).
Comparison of results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance | Month 2
  The results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance) will be compared with data obtained from the first GrossAuTop-1 study (normal pregnancy).
Comparison of results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance | Month 3
  The results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance) will be compared with data obtained from the first GrossAuTop-1 study (normal pregnancy).
Comparison of results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance | Month 4
  The results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance) will be compared with data obtained from the first GrossAuTop-1 study (normal pregnancy).
Comparison of results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance | At delivery
  The results on trophoblastic cell autophagy induction potential, apoptosis and autophagy/apoptosis balance) will be compared with data obtained from the first GrossAuTop-1 study (normal pregnancy).
H.Association between autophagy/apoptosis balance and HbF levels in maternal blood during pregnancy. | Baseline
  Determination of fetal hemoglobin (HbF) in maternal blood, measured in %
H.Association between autophagy/apoptosis balance and HbF levels in maternal blood during pregnancy. | Month 1
  Determination of fetal hemoglobin (HbF) in maternal blood, measured in %
H.Association between autophagy/apoptosis balance and HbF levels in maternal blood during pregnancy. | Month 2
  Determination of fetal hemoglobin (HbF) in maternal blood, measured in %
H.Association between autophagy/apoptosis balance and HbF levels in maternal blood during pregnancy. | Month 3
  Determination of fetal hemoglobin (HbF) in maternal blood, measured in %
H.Association between autophagy/apoptosis balance and HbF levels in maternal blood during pregnancy. | Month 4
  Determination of fetal hemoglobin (HbF) in maternal blood, measured in %
H.Association between autophagy/apoptosis balance and HbF levels in maternal blood during pregnancy. | At delivery
  Determination of fetal hemoglobin (HbF) in maternal blood, measured in %

OTHER OUTCOMES:
I. Constitution of a Biobank | Baseline
  A biobank (plasmabank, serum bank, mononuclear cells) will be set up for ancillary studies on other markers of placental vascular pathologies and venous thromboembolic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Marie PORTES, Dr., Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Mathieu FORTIER, Dr., Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Jean-Christophe GRIS, Pr., Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Eve MOUSTY, Dr., Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Vincent LETOUZEY, Dr., Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Stéphanie HUBERLANT, Dr., Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Chloé BOURGUIGNON, Dr., Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Nimes University Hospital, Nîmes, France